CLINICAL TRIAL: NCT06405646
Title: The Influence of the Concentration of Receptors With Affinity for Cannabidol and Cannabinol on the Risk of Occurrence and Severity of Chronic Orofacial Pain of Muscle Origin
Brief Title: Concentration of Receptors With Affinity for Cannabidiol and Cannabinol and the Effect on Chronic Orofacial Pain of Muscle Origin
Status: Enrolling by invitation | Type: Observational
Sponsor: Wroclaw Medical University (Other)
Responsible Party: Principal Investigator, Joanna Smardz, Investigator, Wroclaw Medical University
Other Study IDs: WMU1/2024
Record Dates: First submitted 2024-05-03; First posted 2024-05-08 (Actual); Last update posted 2025-07-16 (Actual); Status verified 2025-07

CONDITIONS: Myalgia; Muscle Pain; Orofacial Pain; Headache, Tension; Headaches Muscular
Keywords: cannabidiol; cannabinol; TRPV1 receptor; CB1 receptor; CB2 receptor
MeSH Terms: conditions — Myalgia; Facial Pain; Tension-Type Headache

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Study group: Participants with chronic pain in the masticatory muscles
  Interventions: Diagnostic Test: Blood CB1, CB2, TRPV-1 concentration measurement
- Control group: Participants without chronic pain in the masticatory muscles
  Interventions: Diagnostic Test: Blood CB1, CB2, TRPV-1 concentration measurement

INTERVENTIONS:
Diagnostic Test: Blood CB1, CB2, TRPV-1 concentration measurement — In each of the patients blood CB1, CB2, TRPV-1 concentration will be measure

SUMMARY:
The main aim of the presented project will be to examine the concentration of selected receptors (CB1, CB2, TRPV-1) showing affinity for binding to cannabidol (CBD) and cannabinol (CBN) in blood samples collected from people with chronic pain in the masticatory muscles and from people without this pain. Moreover, study participants will be examined by a qualified doctor, according to the validated and standardized international DC/TMD protocol (Diagnostic Criteria for Temporomandibular Disorders) and the criteria included in ICOP-1 (International Classification of Orofacial Pain, 1st edition). The nature and duration of pain, psychoemotional state and central sensitization (the phenomenon of increased reactivity of the nervous system to stimuli) will be determined using validated questionnaires. The obtained results will be subjected to statistical analysis in order to check the relationships between the examined parameters.

DETAILED DESCRIPTION:
Background: Orofacial pain is a common phenomenon in adult patients in Poland. According to available scientific research, it occurs in over half of the population, i.e. 55.9% In its chronic form, orofacial pain may lead to reduced sleep quality, reduced life satisfaction and psychoemotional disorders, including depressive disorders. A popular trend among patients suffering from chronic orofacial pain is the abuse of non-steroidal anti-inflammatory drugs, which in most cases demonstrate low, short-term effectiveness and disproportionate to the side effects. There are scientific reports suggesting that substances such as cannabidol (CBD) and cannabinol (CBN) may be effective in the treatment of chronic nociceptive and neuropathic pain, but there is a clear lack of research on the importance of the concentration of receptors on which they can potentially affect exogenous cannabinoids in the risk of occurrence and development of chronic pain. Of the many receptors to which cannabinoids have affinity, the present study selected those that are involved in neurotransmission related to pain, in particular orofacial pain. The concentrations of CB1, CB2, TRPV-1 receptors will be examined, below is a brief description of each of them to explain their selection.

CB1 and CB2 receptors are G protein-coupled metabotropic receptors and belong to the 7-transmembrane receptor family. CB1 has been detected in central nervous system synapses and sensory neurons. The effect of high CB1 expression in areas closely related to the regulation of pain sensation is the relief of migraine and neuropathic pain. However, CB2 receptors can be found in T and B lymphocytes, spleen, pancreas and tonsils. They work to modulate the release of cytokines and the migration of immune cells in a way that appears to reduce inflammation and some types of pain.

The TRPV-1 receptor is the so-called transient potential 1 vanilloid receptor. They occur primarily at the peripheral endings of nerve fibers, where, as a result of the stimuli that stimulate them, they may participate in the development and conduction of pain. The receptor mediates peripheral pain sensation, able to lower the activation threshold and delay the response of nociceptors. Secondary analgesia following ligand-dependent activation is used in the treatment of some difficult-to-control types of pain, e.g. neuropathic pain. TRPV1 can be activated by endogenous substances, e.g. anandamide, or exogenous substances, e.g. cannabinoids contained in cannabis. It is also worth adding that CBD has the property of blocking FAAH (the enzyme fatty acid amide hydrolase), protecting anandamide against degradation, which means that CBD is also an agonist towards TRPV-1 and protects the natural agonist against degradation by FAAH.

Aim: The aim of this study is to answer how the concentration of the above receptors may influence the occurrence of chronic pain in the masticatory muscles in the study population.

It should be mentioned that CB1, CB2 and TRPV-1 receptors have not yet been included in this research perspective and there are no publications or scientific reports on this subject.

Material and methods:

The study included a study group of 51 people suffering from chronic pain in the masticatory muscles and a control group of 51 healthy people, without pain in the masticatory muscles. Patients will be seen at the Clinic of the University Dental Center in Wrocław. The patient will be qualified based on the standardized and validated international DC/TMD protocol (Diagnostic Criteria for Temporomandibular Disorders) and the criteria included in ICOP-1 (International Classification of Orofacial Pain, 1st edition). The patient's examination will be performed by a qualified dentist.

The control group will include people without chronic pain in the masticatory muscles. The exclusion criteria remain the same as for the study group.

As mentioned above, each study participant will initially undergo an extraoral and intraoral examination based on the validated international DC/TMD (Diagnostic Criteria for Temporomandibular Disorders) protocol. The examinations will be performed by trained dentists.

Patients from both groups will be asked to complete the following validated questionnaires:

* regarding pain - Graded Chronic Pain Scale and McGill Pain Questionnaire
* regarding headache - The Migraine Disability Assessment Test (MIDAS)
* regarding the scale of perceived stress - Perceived Stress Scale - 10 (PSS-10)
* regarding generalized anxiety disorder - Generalized Anxiety Disorder - 7 (GAD-7)
* regarding the scale of somatic symptoms - The Somatic Symptom Scale -8 (SSS8)

The last stage includes collecting a venous blood sample from patients in the study and control groups and determining the concentration of CB1, CB2 and TRPV-1 receptors. The receptors will be determined using specialized ELISA kits.

The collected data will then be subjected to statistical analysis in order to verify the research hypothesis and capture statistically significant relationships.

ELIGIBILITY:
Inclusion Criteria:

* age over 18, under 80
* the presence of chronic pain in the muscles of the masticatory system, which lasts for more than 3 months in accordance with the international criteria included in ICOP-1.

Exclusion Criteria:

* people under 18 years of age
* pregnant or breastfeeding women,
* obese people,
* people with active cancer,
* people with severe systemic diseases, including genetic and neurological diseases,
* people with severe mental illnesses and taking psychoactive substances, people who are taking or have taken antidepressants and/or myorelaxants and/or other drugs that affect neuromuscular activity in the last 12 months
* people addicted to alcohol, drugs and other psychoactive substances
* condition after craniofacial injuries

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with suspicion of Chronic Orofacial Pain of Muscle Origin referred to the Wroclaw Medical University. Healthy controls.
Sampling Method: Probability Sample
Enrollment: 102 (Estimated)
Dates: Start 2025-04-01 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2026-02 (Estimated)

PRIMARY OUTCOMES:
Relationship between the concentration of receptors with affinity for Cannabidol and Cannabinol and the risk of occurrence and severity of chronic orofacial pain of muscle origin | May 5, 2024 - December 31, 2024
  Each participant will undergo blood test focusing on CB1, CB2, TRPV-1 concentration
Assessment of the occurrence of chronic orofacial pain of muscular origin assessed using the Diagnostic Criteria for Temporomandibular Disorders (DC/TMD) protocol. | May 5, 2024 - December 31, 2024
  Each patient will undergo DC/TMD protocol-based clinical examination using DC/TMD examination form assessing incidence of pain of masticatory muscles and surrounding structures.

SECONDARY OUTCOMES:
Assessment of the occurrence of chronic orofacial pain of muscular origin assessed using the Gradual Chronic Pain Scale. | May 5, 2024 - December 31, 2024
  Each participant will fill in Graded Chronic Pain Scale. Scoring Criteria for Grading Chronic Pain Severity: Characteristic Pain Intensity is a 0 to 100 score derived from Questions 1 through 3:Mean (Pain Right Now, Worst Pain, Average Pain) X 10. Disability Score is 0 to 100score derived from Questions 4 through 6:Mean (Daily Activities, Social Activities, Work Activities) X 10. Disability Points: Add the indicated points for Disability Days (Question 7)and for Disability Score. Classification: GRADE 0- No TMD pain in prior 6 months. GRADE I-Low Intensity Characteristic Pain Intensity<50, Low Disability<3 Disability Point. GRADE II -High Intensity Characteristic Pain Intensity >50, LowDisability<3 Disability Points. GRADE III- High Disability3 to 4 Disability Points, Moderately Limiting (Regardless of Characteristic Pain Intensity). GRADE IV- High Disability 5 to 6 Disability Points, Severely Limiting (Regardless of Characteristic Pain Intensity).
Assessment of the occurrence of chronic orofacial pain of muscular origin assessed using the McGill Pain Questionnaire. | May 5, 2024 - December 31, 2024
  Each participant will fill in McGill questionnaire that is composed of 78 words. Respondents choose those that best describe their experience of pain. Scores are tabulated by summing values associated with each word; scores range from 0 (no pain) to 78 (severe pain).
Assessment of the occurrence of chronic orofacial pain of muscular origin assessed using the Migraine Disability Assessment Test (MIDAS) | May 5, 2024 - December 31, 2024
  The Migraine Disability Assessment Test (MIDAS) is a test used by doctors to determine how severely migraines affect a patient's life. Patients are asked questions about the frequency and duration of their headaches, as well as how often these headaches limited their ability to participate in activities at work, at school, or at home.
Assessment of the occurrence of chronic orofacial pain of muscular origin assessed using the Perceived Stress Scale -10 | May 5, 2024 - December 31, 2024
  Each participant will fill in Perceived Stress Scale -10. Scores are obtained by reversing the scores on the four positive items, e.g., 0=4, 1=3, 2=2, etc. and then summing across all 10 items. Items 4,5, 7, and 8 are the positively stated items. It can range from 0 to 40. Scores ranging from 0-13 would be considered low stress,14-26 would be considered moderate stress, 27-40 would be considered high perceived stress.
Assessment of the occurrence of chronic orofacial pain of muscular origin assessed using the Generalized Anxiety Disorder -7 | May 5, 2024 - December 31, 2024
  Each participant will fill in Generalized Anxiety Disorder -7 that consists of 7 items. Total score ranges 0-21 points. Scores of 5, 10, and 15 are taken as the cut-off points for mild, moderate and severe anxiety, respectively.
Assessment of the occurrence of chronic orofacial pain of muscular origin assessed using the Somatic Symptom Scale - 8 | May 5, 2024 - December 31, 2024
  Each participant will fill in the Somatic Symptom Scale - 8 (SSS-8) which is a brief self-report questionnaire used to assess somatic symptom burden. It measures the perceived burden of common somatic symptoms. These symptoms were originally chosen to reflect common symptoms in primary care but they are relevant for a large number of diseases and mental disorders. Scoring: 0-3: no to minimal, 4-7: low, 8-11: medium,12-15: high,16-32: very high.
Assessment of the occurrence of chronic orofacial pain of muscular origin assessed using the Central Sensitizatin Inventory | May 5, 2024 - December 31, 2024
  Each participant will fill in Central Sensitizatin Inventory. This questionnaire consist of two parts. First part includes 25 questions regarding common central sensitivity symptoms. It allows to categorize participant into one of five categories: subclinical (0-29), mild (30-39), moderate (40-49), severe (50-59), and extreme (60-100) Second part is not scored, but it determines if the participant has been diagnosed with certain CSS disorders or related disorders.
Assessment of the occurrence of chronic orofacial pain of muscular origin assessed using the Pain Catastrophizing Scale | May 5, 2024 - December 31, 2024
  Each participant will fill in the Pain Catastrophizing Scale.The Pain Catastrophizing Scale (PCS) will be used to assess pain-related catastrophizing, taking into account items such as exaggeration, hopelessness, and rumination. The PCS consists of 13 items rated on a scale from 0 to 4. The scale can score a maximum of 52 points, with higher scores indicating greater pain-related catastrophic thinking.

CONTACTS AND LOCATIONS:
Locations (1):
- Wroclaw Medical University, Wroclaw, Poland

IPD SHARING:
Plan to Share IPD: Undecided